CLINICAL TRIAL: NCT00373893
Title: Effects of Lidocaine Patch on Intradermal Capsaicin Induced Pain and Hyperalgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 051252
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2005-10

CONDITIONS: Pain; Hyperalgesia
Keywords: Pain; Hyperalgesia; capsaicin
MeSH Terms: conditions — Pain; Hyperalgesia | interventions — Lidocaine

INTERVENTIONS:
Drug: Lidoderm Patch

SUMMARY:
To determine the effects of Lidocaine patch on the pain and hyperalgesia induced by intradermal capsaicin

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo controlled methodology will be conducted. At the session subjects will be exposed to placebo patch and lidocaine patch. Prior to study drug administration, a baseline neurosensory test on the volar aspect of both forearms will be performed and baseline vital signs will be measured. A placebo patch and a lidocaine patch will then be applied to the volar aspect of each forearm. The arms will be randomized to which arm receives placebo and which one receives the lidocaine patch. After four hours of application the right forearm patch will be removed the neurosensory testing will be repeated on the right forearm. After completing the testing, capsaicin (10µl, 10 mg/ml) will be injected intradermally on the volar aspect of the right forearm. Elicited and spontaneous pain scores, blood pressure, heart rate, and respiratory rate will be measured at the time of injection and every 2.5 minutes for 10 minutes. A McGill Pain Questionnaire will be administered at the time of capsaicin injection only. Ten minutes after the capsaicin injection, the hyperalgesic area will be established to von Frey hair, stroking, and heat; the flare response will be outlined; and neurosensory testing will performed halfway between the edge of this defined area and the capsaicin injection site. At the completion of the testing on the right forearm, the left forearm patch will be removed and the procedures described for the right forearm will be repeated for the left forearm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above

Exclusion Criteria:

* Pregnancy.
* Allergy to lidocaine
* Current painful condition
* Current use of analgesics for the treatment of pain
* Lack of ability to understand the experimental protocol and to adequately communicate in English. The neurosensory testing we plan to perform requires the complete cooperation and understanding of the subject. It would be impossible to perform these studies on patients who do not adequately communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-12; Study Completion 2006-02

PRIMARY OUTCOMES:
Neurosensory testing
Four neurosensory tests: warm and cold sensation,warm/cold pain/touch/mechanical pain.
Warm and cold sensation measured w/a Thermal Sensory
Touch will be measured using von Frey hairs. Calibrated von Frey hairs are filaments of varying size. The filament are selected at random and 3 successive stimuli are applied for 1.5 second at 5 second intervals per filament
Mechanical pain will be measured using von Frey hairs. Endpoint will be pain.

SECONDARY OUTCOMES:
Allodynia and Hyperalgesia
At the completion of the stimulation, areas of cutaneous allodynia and hyperalgesia will be mapped. The region of hyperalgesia will be established with a 5.18 von Frey hair, and the area of allodynia with a foam brush gently stroked on the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Wallace, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Center for Pain and Palliative Care, La Jolla, California, United States

REFERENCES:
- [Background] Wallace MS, Laitin S, Licht D, Yaksh TL. Concentration-effect relations for intravenous lidocaine infusions in human volunteers: effects on acute sensory thresholds and capsaicin-evoked hyperpathia. Anesthesiology. 1997 Jun;86(6):1262-72. doi: 10.1097/00000542-199706000-00006. PMID 9197294
- [Background] Wallace MS, Ridgeway B 3rd, Leung A, Schulteis G, Yaksh TL. Concentration-effect relationships for intravenous alfentanil and ketamine infusions in human volunteers: effects on acute thresholds and capsaicin-evoked hyperpathia. J Clin Pharmacol. 2002 Jan;42(1):70-80. doi: 10.1177/0091270002042001008. PMID 11808827
- [Background] Ando K, Wallace MS, Braun J, Schulteis G. Effect of oral mexiletine on capsaicin-induced allodynia and hyperalgesia: a double-blind, placebo-controlled, crossover study. Reg Anesth Pain Med. 2000 Sep-Oct;25(5):468-74. doi: 10.1053/rapm.2000.8584. PMID 11009231
- [Background] Eisenach JC, Hood DD, Curry R, Tong C. Alfentanil, but not amitriptyline, reduces pain, hyperalgesia, and allodynia from intradermal injection of capsaicin in humans. Anesthesiology. 1997 Jun;86(6):1279-87. doi: 10.1097/00000542-199706000-00008. PMID 9197296
- [Background] Eisenach JC, Hood DD, Curry R. Intrathecal, but not intravenous, clonidine reduces experimental thermal or capsaicin-induced pain and hyperalgesia in normal volunteers. Anesth Analg. 1998 Sep;87(3):591-6. doi: 10.1097/00000539-199809000-00018. PMID 9728835
- [Background] Cervero F, Gilbert R, Hammond RGE, Tanner J. Development of secondary hyperalgesia following non-painful thermal stimulation of the skin: a psychophysical study in man. Pain. 1993 Aug;54(2):181-189. doi: 10.1016/0304-3959(93)90207-6. PMID 8233532